CLINICAL TRIAL: NCT04188925
Title: Combined Effect of Laser Acupuncture and Electroacupuncture in Knee Osteoarthritis Patients: a Protocol for a Randomized Controlled Trial
Brief Title: Combined Effect of Laser Acupuncture and Electroacupuncture in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901018A3C501
Record Dates: First submitted 2019-12-01; First posted 2019-12-06 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
Keywords: Electroacupuncture; Laser acupuncture; Low-level laser therapy; Photobiomodulation; Complementary medicine
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sham LA is using the same appearance of LaserPen without energy output to perform the same acupoint as above description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): True LA with EA
  Interventions: Device: Laser Acupuncture
- Group B (Sham Comparator): Sham LA with EA
  Interventions: Device: Sham Laser Acupuncture

INTERVENTIONS:
Device: Laser Acupuncture — The LA is using a gallium aluminum arsenide LaserPen (maximal power, 150 mW; wavelength, 810nm; area of probe, 0.03cm2; power density, 5W/cm2; pulsed wave; RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany). The LA treatment will be applied to EX-LE5, ST35, and BL40 for 80 seconds, under power 150mW, to deliver a total treatment dose of 6 Joule/ cm2.
  The EA is the combination of acupuncture and transcutaneous electrical nerve stimulator. The transcutaneous electrical nerve stimulator is produced by Ching Ming Medical Device Company. This machine is verified by Department of Health in Taiwan, with the ID number 001147. We perform acupuncture on GB33, GB34, SP9, SP10, and ST36.
  Arms: Group A
Device: Sham Laser Acupuncture — Sham LA is using the same appearance of LaserPen without energy output to perform the same acupoint as above description. Both of the LaserPen in two groups are labeled with A and B, one of them is revised by the company to become the sham LA. The outward of both LaserPen are the same and our physician does not know which one is the real.
  Arms: Group B

SUMMARY:
Background:

Knee osteoarthritis (KOA) is a common degenerative joint disorder affected 250 million people globally. It can not only result in disability, but also associated with cardiovascular disease and mortality. The most common treatment for KOA is non-steroidal anti-inflammatory drug. However, the effect of analgesic is limited and may complicate with side effect. Hence, many patients search for complementary and alternative medicine. Acupuncture is one of the most popular complementary treatment with good analgesic effect and less side effect. Electroacupuncture (EA) or laser acupuncture (LA) was reported effective in pain control in knee osteoarthritis patients. However, there is no study about combination effect of EA and LA.

Methods:

This protocol is a randomized controlled trial investigating the combination effect of EA and LA on KOA. Fifty participants diagnosed KOA with aged more than 50 years old and knee pain more than 3 months were recruited and randomly assigned to the experimental group (EA plus LA) or sham group (EA plus LA without laser output) in clinical research center. The subjects will undergo EA plus LA treatment thrice a weeks for 4 weeks. The experimental group will receive acupuncture at GB33, GB34, SP9, SP10, and ST36 with transcutaneous electrical nerve stimulator on the GB34+33 and SP9+10., and the LA deliver 6 Joule of energy at EX-LE5, ST35, and BL40. The subjects in sham group will receive the same way but the LA is without any laser output. Outcome measurement will include visual analogue scale (VAS), Western Ontario McMaster Universities Osteoarthritis Index (WOMAC), Knee injury and osteoarthritis outcome (KOOS), body composition analysis, knee range of motion test, muscle stiffness test, standing on one foot test, and the 30-second chair stand test before intervention and after 4 weeks intervention. The result will be analyze and compared between the experimental group and sham group using the paired t test and one-way analysis of variance.

Objectives:

The aim of this protocol is to investigate the combination effect of EA and LA in KOA patients.

ELIGIBILITY:
Inclusion Criteria:

* VAS more than 3 point when daily activity
* Kellgren-Lawrence Grading Scale grade 1 to 3 on knee X-ray
* Provided informed consent

Exclusion Criteria:

* History of knee arthroplasty, traumatic injury related joint deformity,
* Body mass index more than 35
* pacemaker insertion, photosensitivity
* who had undergone intra-articular injection or acupuncture in recent one month
* other factors that may affect the evaluation of the outcome, such as psychiatric disorder or moderate mental retardation etc.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analog Score | Through study completion, an average of 4 weeks
  Visual Analog Score for pain during activity; change from baseline at 4 weeks; scoring from 0 to 10, and the higher scores indicate the worse condition
Use of analgesics | Through study completion, an average of 4 weeks
  Frequency of analgesics

SECONDARY OUTCOMES:
Change of the score of Western Ontario and McMaster Universities Arthritis Index | Through study completion, an average of 4 weeks
  Questionnaires for the function in patients with OA knee; change from baseline at 4 weeks; scoring from 0 to 68, and the higher scores indicate the worse condition
Change of the percentage of Knee Injury and Osteoarthritis Outcome Score | Through study completion, an average of 4 weeks
  Questionnaires for the function in patients with OA knee; change from baseline at 4 weeks; scoring from 0 to 100 percentage, and the higher percentage indicates the better condition
Change of the muscle stiffness of quadriceps | Through study completion, an average of 4 weeks
  The value is measured by Myoton Digital Palpation Device; change from baseline at 4 weeks
Change of the angle of knee range of motion | Through study completion, an average of 4 weeks
  The range between flexion and extension of the knee; change from baseline at 4 weeks
Change of the minutes of standing on one foot test | Through study completion, an average of 4 weeks
  The patient stands on one foot with hands on hips and eye opening. The time that the patient can stand on one foot was recorded; change from baseline at 4 weeks
Change of the times of 30-second chair stand test | Through study completion, an average of 4 weeks
  The patient sits on the chair with bilateral feet stepping on the ground and hands cross beyond chest. Then he/she stands up and then sits down. The definition of once is completing one standing up and then sitting down. The number of times that the patient could stand up and then sit down within 30 seconds; change from baseline at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No